CLINICAL TRIAL: NCT01202188
Title: A 26-week Treatment Multi-center, Randomized, Double-blind, Parallel-group, Placebo and Active Controlled (Open Label) Study to Assess the Efficacy, Safety and Tolerability of QVA149 (110/50 μg q.d.) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of Once-daily (q.d.) QVA149 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2303; 2009-017772-25 (EudraCT Number)
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: QVA149, COPD, combination bronchodilator, indacaterol, glycopyrronium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate; indacaterol-glycopyrronium combination; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- indacaterol and glycopyrronium (QVA149) (Experimental): QVA149 110/50 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDPPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
  Interventions: Drug: indacaterol and glycopyrronium (QVA149)
- glycopyrronium (NVA237) (Active Comparator): NVA237 50 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDDPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
  Interventions: Drug: glycopyrronium (NVA237)
- indacaterol (QAB149) (Active Comparator): QAB149 150 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDDPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
  Interventions: Drug: indacaterol (QAB149)
- tiotropium (Active Comparator): Tiotropium 18 μg capsules for inhalation delivered once daily via HandiHaler® device for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
  Interventions: Drug: tiotropium
- Placebo (Placebo Comparator): Matching placebo capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDDPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indacaterol and glycopyrronium (QVA149) — Capsules for inhalation delivered via SDDPI.
  Arms: indacaterol and glycopyrronium (QVA149)
Drug: glycopyrronium (NVA237) — Capsules for inhalation delivered via SDDPI.
  Arms: glycopyrronium (NVA237)
Drug: indacaterol (QAB149) — Capsules for inhalation delivered via SDDPI.
  Arms: indacaterol (QAB149)
Drug: tiotropium — Capsules for inhalation delivered via HandiHaler® device.
  Arms: tiotropium
Drug: placebo — Placebo to match capsules for inhalation delivered via SDDPI.
  Arms: Placebo

SUMMARY:
The purpose of this study is to provide pivotal efficacy and safety data for QVA149 in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 yrs
* Smoking history of at least 10 pack years
* Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2008)
* Post-bronchodilator FEV1 < 80% and ≥ 30% of the predicted normal value and post-bronchodilator FEV1/FVC (forced vital capacity) <70%

Exclusion Criteria:

* Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for inhaled anticholinergic agents and β2 agonists
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2144 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (166):
- United States (14):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Johnson City, Tennessee
- Australia (5):
  - Novartis Investigative Site, Daw Park
  - Novartis Investigative Site, Glebe
  - Novartis Investigative Site, Kogarah
  - Novartis Investigative Site, Nedlands
  - Novartis Investigative site, New Lambton
- Bulgaria (5):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
- Canada (7):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Courtice, Ontario
  - Novartis Investigative Site, Mississuaga, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (4):
  - Novartis Investigative Site, Beuvry
  - Novartis Investigative Site, Bourges
  - Novartis Investigative Site, Ferolles-Attily
  - Novartis Investigative Site, Rennes
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Geesthacht
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Witten
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (6):
  - Novartis INvestigative Site, Balassagyarmat
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Tatabánya
- Japan (33):
  - Novartis Investigative Site, Asahikawa
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Chūōku
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hachiōji
  - Novartis Investigative Site, Hamakita
  - Novartis Investigative Site, Himeji
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Hitachi
  - Novartis Inverstigative Site, Iwata
  - Novartis Investigative Site, Kamogawa
  - Novartis Investigative Site, Kishiwada
  - Novartis Investigative Site, Kiyose
  - Novartis Investigative Site, Kurashiki
  - Novartis Investigative Site, Matsumoto
  - Novartis Investigative Site, Matsusaka
  - Novartis Investigative Site, Minatoku
  - Novartis Investigative Site, Moriya
  - Novartis Investigative Site, Nagaoka
  - Novartis Investigative Site, Nagoya
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Obihiro
  - Novartis Investigative Site, Sakai
  - Novartis Investigative Site, Sakaidechō
  - Novartis Investigative Site, Sapporo
  - Novartis Investigative Site, tabashi City
  - Novartis Investigative Site, Tachikawa
  - Novartis Investigative Site, Takatsuki
  - Novartis Investigative Site, Tsu
  - Novartis Investigative Site, Yabu
  - Novartis Investigative Site, Yanagawa
  - Novartis Investigative Site, Yatsushiro
  - Novartis Investigative Site, Yonezawa
- Philippines (5):
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Pasay
  - Novartis Investigative Site, Quezon City
- Poland (4):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Proszowice
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Warsaw
- Russia (9):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Nizhny Novogorod
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Ufa
- Slovakia (12):
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bojnice
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Humenné
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Liptovský Hrádok
  - Novartis Investigative Site, Partizánske
  - Novartis Investigative Site, Prievidza
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Trstená
  - Novartis Investigative Site, Zvolen
  - Novartis Investigative Site, Žilina
- South Africa (5):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Lyttleton
  - Novartis Investigative Site, Pretoria
- Spain (19):
  - Novartis Investigative Site, Alzira
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Canet de Mar
  - Novartis Investigative Site, Centelles
  - Novartis Investigative Site, Ferrol
  - Novartis Investigative Site, Fuenlabrada
  - Novartis Investigative Site, les Borges del Camp
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Mataró
  - Novartis Investigative Site, Mérida
  - Novartis Investigative Site, Motril
  - Novartis Investigative Site, Móstoles
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Ponferrada
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Salt
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Vic
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Münchenstein
  - Novartis Investigative Site, Neuchâtel
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Chai-Yi
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (11):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Bolu
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Çanakkale
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Manisa
  - Novartis Investigative Site, Mersin
- United Kingdom (10):
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cambs
  - Novartis Investigative Site, Chelmsford
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Herts
  - Novartis Investigative Site, Isle of Wight
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Kulich K, Keininger DL, Tiplady B, Banerji D. Symptoms and impact of COPD assessed by an electronic diary in patients with moderate-to-severe COPD: psychometric results from the SHINE study. Int J Chron Obstruct Pulmon Dis. 2015 Jan 7;10:79-94. doi: 10.2147/COPD.S73092. eCollection 2015. PMID 25609942

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 14 day run-in period prior to randomization.
Groups:
- Indacaterol and Glycopyrronium (QVA149): QVA149 110/50 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDDPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
- Glycopyrronium (NVA237): NVA237 50 μg capsules for inhalation delivered once daily via a single-dose dry powder inhaler (SDDPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and salbutamol/albuterol was available for use as rescue medication throughout the study.
Period: Overall Study
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Started | 475 | 477 | 475 | 483 | 234
Safety Set; Received Study Drug | 474 | 476 | 473 | 480 | 232
Completed | 437 | 421 | 422 | 441 | 189
Not Completed | 38 | 56 | 53 | 42 | 45
Not completed — Protocol deviation | 14 | 8 | 12 | 10 | 11
Not completed — Subject withdrew consent | 12 | 13 | 22 | 11 | 13
Not completed — Adverse Event | 5 | 23 | 13 | 10 | 10
Not completed — Administrative problems | 3 | 2 | 1 | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 2 | 8 | 2 | 5 | 8
Not completed — Lost to Follow-up | 1 | 1 | 0 | 4 | 1
Not completed — Death | 1 | 1 | 1 | 1 | 0
Not completed — Abnormal test procedure result (s) | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Safety Set that includes all participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo | Total
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232 | 2135
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.88) | 63.6 (8.78) | 64.3 (9.04) | 63.5 (8.73) | 64.4 (8.58) | 63.9 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 122 | 108 | 120 | 63 | 525
  Male | 362 | 354 | 365 | 360 | 169 | 1610

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume In One Second (FEV1) After 26 Weeks of Treatment
Description: Spirometry was performed according to internationally accepted standards. Trough FEV1 was defined as the mean of the 23 hour 15 minute and 23 hour 45 minute post-dose values. A mixed model was used with treatment as a fixed effect with baseline FEV1 and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 23 hours 15 minutes and 23 hour 45 minute post-dose Week 26
Population: Participants from the Full Analysis Set, defined as all randomized participants who received at least one dose of study drug, with data available for analysis. Data was imputed with last observation carried forward. Data within 6 hours of rescue medication use or 7 days of systemic corticosteroid use is excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol and Glycopyrronium (QVA149): QVA149 110/50 μg capsules for inhalation delivered once daily via a single-dose dry powder inhaler (SDPPI) for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and Salbutamol/albuterol was available for use as rescue medication throughout the study.
- Indacaterol (QAB149): QAB149 150 μg capsules for inhalation delivered once daily via a SDDPI for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and Salbutamol/albuterol was available for use as rescue medication throughout the study.
- Glycopyrronium (NVA237): NVA237 50 μg capsules for inhalation delivered once daily via a SDDPI for 26 weeks.Participants remained on a stable dose of inhaled corticosteroid (ICS) and Salbutamol/albuterol was available for use as rescue medication throughout the study.
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237)
Number analyzed (Participants) | 442 | 435 | 424
Liters | 1.45 (0.010) | 1.38 (0.010) | 1.36 (0.010)

2. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score at Week 26
Description: A trained assessor interviewed the patient and graded the degree of impairment due to dyspnea (difficulty breathing). TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score. A mixed model was used with treatment as a fixed effect with Baseline Dyspnea Index Score and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: Week 26
Population: Participants from the Full Analysis Set, included all participants who received at least one dose of study drug, with data available for analysis. Missing data were imputed with Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Placebo: Matching Placebo capsules for inhalation delivered once daily via a SDDPI for 26 weeks. Participants remained on a stable dose of inhaled corticosteroid (ICS) and Salbutamol/albuterol was available for use as rescue medication throughout the study.
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Placebo
Number analyzed (Participants) | 439 | 193
Score on a scale | 2.72 (0.170) | 1.63 (0.230)

3. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 26
Description: SGRQ is a health related quality of life questionnaire consisting of 51 items in three areas: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). The total score is 0 to 100 with a higher score indicating poorer health status. A mixed model was used with treatment as a fixed effect with Baseline SGRQ and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 26 weeks
Population: Participants from the Full Analysis Set,included all participants who received at least one dose of study drug, with data available for analysis. Missing data were imputed with Last Observation Carried Forward but not more than 14 weeks and data within 4 weeks of day 1 were not carried forward.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Placebo
Number analyzed (Participants) | 441 | 196
Score on a scale | 37.01 (0.679) | 40.02 (0.941)

4. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication Over 26 Weeks
Description: The number of puffs of rescue medication taken in the previous 12 hours was record in patient diary in the morning and in the evening for 26 weeks. The total number of puffs per day was calculated and divided by the number of days with data to determine the mean daily number of puffs of rescue medication for each patient. Rescue medication data recorded during the 14 day run-in was used to calculate the baseline. A negative change from baseline indicates improvement. A mixed model was used with treatment as a fixed effect with baseline number of puffs and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: Baseline, Week 26
Population: Participants from the full analysis, consisting of all randomized participant who received study drug, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Placebo
Number analyzed (Participants) | 419 | 199
Puffs per day | -1.88 (0.105) | -0.92 (0.147)

5. Secondary Outcome: Trough Forced Expiratory Volume In One Second (FEV1) After 26 Weeks of Treatment With QVA149, QAB149 and NVA237 Compared to Placebo
Description: as for outcome 1
Time Frame: 23 hours 15 minutes and 23 hour 45 minute post-dose Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Placebo
Number analyzed (Participants) | 442 | 435 | 424 | 191
Liters | 1.45 (0.010) | 1.38 (0.010) | 1.36 (0.010) | 1.25 (0.015)

6. Secondary Outcome: Trough Forced Expiratory Volume In One Second (FEV1) After 26 Weeks of Treatment With QVA149 Compared to Tiotropium
Description: as for outcome 1
Time Frame: 23 hours 15 minutes and 23 hour 45 minute post-dose Week 26
Population: Participants from the Per-protocol Set, randomized participants who received at least one dose of study drug without major protocol deviations. Data was imputed with last observation carried forward. Data within 6 hours of rescue medication use or 7 days of systemic corticosteroid use is excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Tiotropium: Tiotropium 18 μg capsules for inhalation delivered once daily via the manufacturer's proprietary device for 26 weeks.Participants remained on a stable dose of inhaled corticosteroid (ICS) and Salbutamol/albuterol was available for use as rescue medication throughout the study.
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 387 | 382
Liters | 1.46 (0.011) | 1.39 (0.011)

7. Secondary Outcome: Baseline Transitional Dyspnea Index (BDI/TDI) Focal Score at Week 12 and Week 26
Description: A trained assessor interviewed the patient and graded the degree of impairment due to dyspnea (difficulty breathing). BDI/TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. BDI was measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best). TDI captures changes from baseline. Each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score.
  A mixed model was used with treatment as a fixed effect with Baseline Dyspnea Index Score and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators as covariates and included baseline smoking status, baseline inhaled corticosteroids and region as fixed effects with center nested within region as a random effect.
Time Frame: Baseline, Week 12, Week 26
Population: Participants from the Full Analysis Set, included all participants who received at least one dose of study drug, with data available for analysis. Missing data were imputed with Last Observation Carried Forward but not more than 14 weeks and data within 4 weeks of day 1 were not carried forward.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 442 | 443 | 435 | 445 | 200
Score on a scale
  BDI_ baseline for Week 12 | 6.45 (0.100) | 6.28 (0.096) | 6.21 (0.097) | 6.43 (0.094) | 6.53 (0.154)
  TDI Week 12 | 2.44 (0.158) | 2.18 (0.157) | 2.04 (0.158) | 1.81 (0.158) | 1.22 (0.215)
  BDI_baseline for Week 26 (n=439,440,424,441,193) | 6.45 (0.101) | 6.28 (0.097) | 6.22 (0.097) | 6.46 (0.095) | 6.56 (0.157)
  TDI Week 26 (n=439,440,424,441,193) | 2.72 (0.170) | 2.47 (0.171) | 2.52 (0.172) | 2.21 (0.171) | 1.63 (0.230)

8. Secondary Outcome: Percentage of Patients With a Clinically Important Improvement of at Least 1 Point in TDI Focal Score After 26 Weeks of Treatment
Description: A trained assessor interviewed the patient and graded the degree of impairment due to dyspnea (difficulty breathing) at Week 12 and Week 26. TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. The BDI (baseline) was measured at Day 1. The TDI captures changes from baseline. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Percentage of participants | 68.1 | 64.6 | 63.7 | 59.2 | 57.5

9. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score After 12 and 26 Weeks of Treatment
Description: as for outcome 3
Time Frame: Week 12, Week 26
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 448 | 446 | 441 | 454 | 205
Score on a scale
  12 Weeks | 37.56 (0.659) | 38.55 (0.662) | 39.40 (0.663) | 39.94 (0.658) | 41.55 (0.900)
  26 Weeks (n=441,443,430,450,196) | 37.01 (0.679) | 38.10 (0.680) | 38.19 (0.686) | 39.14 (0.677) | 40.02 (0.941)

10. Secondary Outcome: Percentage of Patients With a Clinically Important Improvement From Baseline of at Least 4 Units in the SGRQ Total Score After 26 Weeks of Treatment
Description: SGRQ is a health related quality of life questionnaire consisting of 51 items in three areas: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). The total score is 0 to 100 with a higher score indicating poorer health status.
Time Frame: Baseline, Week 26
Population: Participants from the Full Analysis Set, that included all participants who received at least one dose of study drug, with data available for analysis. Missing data were imputed with Last Observation Carried Forward but not more than 14 weeks and data within 4 weeks of day 1 were not carried forward.
Measure: Number; unit: Percentage of participants
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Percentage of participants | 63.7 | 63.0 | 60.5 | 56.4 | 56.6

11. Secondary Outcome: Percentage of Nights With "No Night Time Awakenings" Over 26 Weeks
Description: A day with no night time awakenings is defined from the diary data as any day where the patient did not wake up due to COPD symptoms. The percentage of nights is calculated by the number of days with no nighttime awakenings/total number of days with evaluable data X 100. A mixed model was used with treatment as a fixed effect with baseline Percent days and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 26 Weeks
Population: Participants from the Full Analysis Set, all randomized participants who received study drug, with evaluable diary data (at least 40 days) for analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 418 | 413 | 399 | 422 | 198
Percentage of nights | 63.68 (1.473) | 62.48 (1.479) | 58.64 (1.500) | 60.00 (1.469) | 53.67 (2.047)

12. Secondary Outcome: Percentage of Days With "No Daytime Symptoms" Over 26 Weeks
Description: A day with no day time symptoms is defined from the diary data as any day where the patient recorded no coughing, no wheezing, no sputum production and no breathlessness during the previous 12 hours (approximately 8AM to 8PM). The percentage of days is calculated by the number of days with no daytime symptoms/total number of days with evaluable data X 100. A mixed model was used with treatment as a fixed effect with baseline Percent of days and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 26 Weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 415 | 410 | 395 | 418 | 195
Percentage of days | 7.49 (0.931) | 9.17 (0.933) | 6.40 (0.948) | 5.54 (0.928) | 4.44 (1.294)

13. Secondary Outcome: Percentage of "Days Able to Perform Usual Daily Activities" Over 26 Weeks
Description: Patients answered the question "Did your respiratory symptoms stop you performing your usual activities today?-Not at all in their daily diary. The percentage of days is calculated by the number of days patient is able to perform daily activities/total number of days with evaluable data X 100. A mixed model was used with treatment as a fixed effect with baseline Percent of Days and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 26 Weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 415 | 410 | 395 | 418 | 195
Percentage of days | 45.97 (1.578) | 40.94 (1.582) | 40.10 (1.607) | 37.52 (1.572) | 34.49 (2.197)

14. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication at Week 12 and Week 26
Description: as for outcome 4
Time Frame: Baseline, Week 12, Week 26
Population: Participants from the full analysis, consisting of all randomized participant who received study drug, with data available for analysis at Week 12 and Week 26.
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 420 | 420 | 413 | 427 | 203
Puffs per day
  Change from Baseline (BL) at Week 12 | -1.82 (0.102) | -1.46 (0.102) | -1.22 (0.103) | -1.28 (0.102) | -0.83 (0.141)
  Change from BL at Week 26 (n=419,416,403,424,199) | -1.88 (0.105) | -1.57 (0.106) | -1.22 (0.107) | -1.34 (0.105) | -0.92 (0.147)

15. Secondary Outcome: Change From Baseline (BL) in the Daytime and Night Time Rescue Medication Use (Number of Puffs) Over 26 Weeks
Description: The number of puffs of rescue medication taken in the previous 12 hours was record in patient diary in the morning and in the evening for 26 weeks. The total number of puffs in the morning and evening were calculated and divided by the number of days with data to determine the mean daily number of daytime and nighttime puffs. A mixed model was used with treatment as a fixed effect with baseline number of puffs and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline (BL) ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Puffs
  Daytime Change from BL (n=415,410,395,418,195) | -1.11 (0.061) | -0.96 (0.062) | -0.75 (0.063) | -0.83 (0.061) | -0.58 (0.086)
  Nighttime Change from BL (n=418,413,399,422,198) | -0.78 (0.049) | -0.63 (0.049) | -0.48 (0.050) | -0.52 (0.049) | -0.34 (0.069)

16. Secondary Outcome: Percentage of "Days With no Rescue Medication Use" Over 26 Weeks
Description: A day with no rescue medication use is defined from the diary data as any day where the patient recorded no rescue medicine use during the previous 12 hours. The percentage of days is calculated by the number of days with no rescue medicine use/total number of days with evaluable data X 100. A mixed model was used with treatment as a fixed effect with baseline number of puffs and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: 26 Weeks
Population: Participants from the full analysis set (all randomized participants who received at least one dose of study drug) with evaluable data (at least 40 days of diary data) available for analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 418 | 411 | 397 | 419 | 196
Percentage of days | 47.09 (1.752) | 44.81 (1.764) | 37.74 (1.790) | 36.51 (1.752) | 34.76 (2.437)

17. Secondary Outcome: Standardized FEV1 (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours at Day 1 and Week 26
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. A mixed model was used with treatment as a fixed effect with baseline FEV1 and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: From 5 minutes to 4 hours post-dose Day 1 and Week 26
Population: Participants from full analysis set, all randomized participants who received study drug, with data available for analysis. Data within 6 hours of rescue medication use or 7 days of systemic corticosteroid use is excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 464 | 471 | 464 | 473 | 228
Liters
  Day 1 | 1.52 (0.006) | 1.46 (0.006) | 1.49 (0.006) | 1.44 (0.006) | 1.30 (0.008)
  Week 26 (n=433,418,412,435,186) | 1.57 (0.010) | 1.46 (0.010) | 1.43 (0.010) | 1.44 (0.010) | 1.23 (0.015)

18. Secondary Outcome: Standardized FEV1 (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 12 Hours at Day 1 and Week 26
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 4, 8, 12 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. A mixed model was used with treatment as a fixed effect with baseline FEV1 and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: From 5 minutes to 12 hours post-dose Day 1 and Week 26
Population: Participants from the 24 hour serial spirometry subset of the full analysis set (all randomized participants who received study drug) with data available for analysis. Data within 6 hours of rescue medication use or 7 days of systemic corticosteroid use is excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 64 | 64 | 63 | 70 | 31
Liters
  Day1 | 1.50 (0.017) | 1.40 (0.017) | 1.42 (0.018) | 1.38 (0.017) | 1.24 (0.023)
  Week 26 (n=60,55,58,67,27) | 1.52 (0.027) | 1.39 (0.027) | 1.39 (0.028) | 1.39 (0.027) | 1.18 (0.036)

19. Secondary Outcome: Standardized FEV1 (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 23 Hours 45 Minutes at Week 26
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 4, 8, 12, 23 hours 15 minutes and 23 hours 45 minutes post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. A mixed model was used with treatment as a fixed effect with baseline FEV1 and FEV1 prior to inhalation and FEV1 60 minutes post inhalation of two short acting bronchodilators (components of reversibility at Day -14) as covariates. The model also included baseline smoking status (current/ex-smoker), baseline ICS use (Yes/No) and region as fixed effects with center nested within region as a random effect.
Time Frame: From 5 minutes to 23 hours 45 minutes post-dose Week 26
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 60 | 55 | 58 | 67 | 27
Liters | 1.46 (0.026) | 1.35 (0.027) | 1.35 (0.027) | 1.36 (0.026) | 1.15 (0.036)

20. Secondary Outcome: 24 Hour Holter Monitoring in a Subset of Patients
Description: 24-hourly mean heart rate was performed using a Holter Monitor at Weeks 12 and 26 in a subgroup of patients. Mixed model: heart rate = treatment + baseline heart rate + baseline smoking status + baseline ICS use + region + center (region) + error. Center was included as a random effect nested within region.
  The 24-hourly mean heart rate is the mean heart rate over the 24 hour period, derived using hourly mean heart rate beats per minute.
Time Frame: Week 12, Week 26
Population: Safety Set Holter Group-a subset of the Safety participants that included all randomized participants who received at least one dose of study drug and participated in the 24 hour Holter monitoring with evaluable data available for analysis. No participants in the Titotropium arm participated in the Holter Monitoring.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Placebo
Number analyzed (Participants) | 59 | 52 | 55 | 24
beats per minute
  Week 12 (n=35,38,27,15) | 80.8 (1.5) | 79.9 (1.35) | 79.4 (1.57) | 78.9 (1.95)
  Week 26 (n=36,36,26,16) | 79.8 (1.68) | 78.6 (1.57) | 80.5 (1.75) | 77.0 (2.09)

21. Secondary Outcome: Rate of Moderate or Severe COPD Exacerbation
Description: Rate of moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Time Frame: 26 Weeks
Measure: Number; unit: Exacerbations per year
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Exacerbations per year | 0.46 | 0.59 | 0.52 | 0.45 | 0.75

22. Secondary Outcome: Percentage of Patients With at Least One Moderate or Severe COPD Exacerbation Over the 26 Week Treatment Period
Time Frame: 26 Weeks
Population: Full Analysis Set includes all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Percentage of participants | 17.9 | 21.6 | 18.8 | 17.7 | 25.8

23. Secondary Outcome: Percentage of Participants With COPD Exacerbations Requiring Hospitalization or Treatment With Systemic Corticosteroids and/or Antibiotics But no Hospitalization
Time Frame: 26 Weeks
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Number analyzed (Participants) | 474 | 476 | 473 | 480 | 232
Percentage of participants
  Requiring hospitalization | 2.1 | 2.5 | 1.9 | 1.0 | 3.0
  Corticosteroids_Antibiotics-No hospitalization | 16.7 | 19.7 | 17.8 | 16.9 | 23.3

ADVERSE EVENTS:
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Indacaterol (QAB149) | Glycopyrronium (NVA237) | Tiotropium | Placebo
Serious Adverse Events (participants affected / at risk) | 22/474 | 26/476 | 29/473 | 19/480 | 13/232
Other Adverse Events (participants affected / at risk) | 166/474 | 189/476 | 185/473 | 172/480 | 102/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium (QVA149) (N=474) | Indacaterol (QAB149) (N=476) | Glycopyrronium (NVA237) (N=473) | Tiotropium (N=480) | Placebo (N=232)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 3 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Moraxella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 3 | 3 | 3
Respiratory tract infection bacterial (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 9 | 7 | 7
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium (QVA149) (N=474) | Indacaterol (QAB149) (N=476) | Glycopyrronium (NVA237) (N=473) | Tiotropium (N=480) | Placebo (N=232)
Nasopharyngitis (Infections and infestations) | 31 | 35 | 46 | 40 | 23
Upper respiratory tract infection (Infections and infestations) | 20 | 31 | 20 | 24 | 13
Upper respiratory tract infection bacterial (Infections and infestations) | 10 | 12 | 15 | 22 | 13
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 131 | 144 | 146 | 133 | 87
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 38 | 18 | 21 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.